CLINICAL TRIAL: NCT04085198
Title: Light Physics Enhanced Camera Navigation in No-touch Hysteroscopy: Randomized Controlled Trial
Brief Title: Light Physics Enhanced Camera Navigation in Hysteroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Huseyin Kiyak, Principal Investigator, M.D., Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Huseyin5
Record Dates: First submitted 2019-09-09; First posted 2019-09-11 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No-touch technique with the application of light physics rules (Active Comparator): This procedure will be performed by the gynecologists who are familiar to the rules of the 'lights physics' and are currently 'lights physics' rules in their clinical practice. The brightness or darkness of the tissue which reflects the distance between the light source and the surrounding tissue will be used to find the correct route from the vagina introitus to the uterine cavity.
  Interventions: Procedure: Light physics enhanced 'no-touch' hysteroscopy
- Control (Placebo Comparator): Patients in this arm of the study protocol will receive standard hysteroscopy with 'no-touch' technique without the utilization of the 'lights physics' rules. The gynecologist performing this procedure will find their route from the vagina introitus to the uterine cavity by the identification of the anatomical structures on their way.
  Interventions: Procedure: Standard hysteroscopy

INTERVENTIONS:
Procedure: Light physics enhanced 'no-touch' hysteroscopy — The light source used in hysteroscopy provides an illumined environment during the imagination with these techniques. During hysteroscopy, the light reflecting from the adjacent tissue appears bright, however, this reflection is weaker in farther tissue and these structures appear dark. This information will be used in determining the route from the vaginal introitus to the uterine cavity during the hysteroscopy.
  Arms: No-touch technique with the application of light physics rules
Procedure: Standard hysteroscopy — Anatomical structures as illumined by the light source of the camera will be used to find the route from the vaginal introitus to the uterine cavity
  Arms: Control

SUMMARY:
Office hysteroscopy is the gold standard technique in the diagnosis of the intrauterine pathologies. Some interventions may also be carried out through the hysteroscopy. No-touch hysteroscopy technique confers several advantages in terms of patient discomfort over the traditional technique. Clinicians performing the hysteroscopy find their way from the vaginal introitus to the uterine cavity through direct visualization of the anatomic structures on their route. The investigators hypothesize that the utilization of the information derived from the 'light physics' would facilitate camera navigation during no-touch hysteroscopy and consequently ease reaching the uterus. This study aimed to compare the standard no-touch technique with the 'light physics' enhanced camera navigation in terms of patient comfort and procedural pain.

DETAILED DESCRIPTION:
Office hysteroscopy is basically used in the diagnosis of the intrauterine pathologies. 'No touch' vaginal hysteroscopy does not require a speculum or tenaculum; thus, confers advantages in terms of patient discomfort over the traditional technique. The source of the pain in traditional hysteroscopy is the distention of the uterine cavity with the saline and the contact of the hysteroscopy equipment with the vagina and the cervical canal. The benefit in the pain obtained with the 'no-touch' technique is derived from the limitation of the contact of the hysteroscopy equipment with the vagina and the cervical canal. Clinicians performing the hysteroscopy find their way from the vaginal introitus to the uterine cavity through direct visualization of the anatomic structures on their route.

Physics has been critical in the development of endoscopic techniques such as laparoscopy, cystoscopy, and hysteroscopy. The light source provides an illumined environment during the imagination with these techniques. During hysteroscopy, the light reflecting from the adjacent tissue appears bright, however, this reflection is weaker in farther tissue and these structures appear dark. With this in mind, the investigators hypothesize that the utilization of the information derived from the 'light physics' would facilitate camera navigation during no-touch hysteroscopy and consequently ease reaching the uterus. This study aimed to compare the standard no-touch technique with the 'light physics' enhanced camera navigation in terms of patient comfort and procedural pain.

ELIGIBILITY:
Inclusion Criteria:

* Must be scheduled for No-touch Office hysteroscopy procedure with a diagnostic purpose
* Must be nulliparous

Exclusion Criteria:

* Multiparous women
* Previous cesarean section
* Cervical stenosis

Ages: 20 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2019-09-13 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
Procedural Pain | immediately after the procedure
  The visual analogue scale score for procedural pain (0 to 10, 10 as the most painful)
Procedure time | procedure
  The time required to perform the hysteroscopy

SECONDARY OUTCOMES:
Patient satisfaction | immediately after the procedure
  Patients' self-reported satisfaction (satisfied or not satisfied with the procedure)

CONTACTS AND LOCATIONS:
Overall Officials: Huseyin Kiyak, MD, Principal Investigator — University of Health Sciences, Faculty of Medicine
Locations (1):
- Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Please Enter the State Or Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No